CLINICAL TRIAL: NCT04583683
Title: Effects of Very Low Calorie Diet vs Metabolic Surgery on Weight Loss and Obesity Comorbidities: a Randomized Controlled Trial
Brief Title: Effects of Very Low Calorie Diet vs Metabolic Surgery on Weight Loss and Obesity Comorbidities
Acronym: ARGOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20203009
Record Dates: First submitted 2020-09-30; First posted 2020-10-12 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Obesity, Morbid; Obesity; Diet, Healthy; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Dietary Supplements; Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive lifestyle modification: Very low calorie diet (Active Comparator): Patients will undergo a very low calorie diet
  Interventions: Behavioral: Very low calorie diet with Fortimel (Nutricia) supplementation
- Metabolic Surgery (Active Comparator): Patients will undergo metabolic surgery
  Interventions: Procedure: Metabolic Surgery

INTERVENTIONS:
Behavioral: Very low calorie diet with Fortimel (Nutricia) supplementation — Patients will undergo a very low calorie diet
  Arms: Intensive lifestyle modification: Very low calorie diet
Procedure: Metabolic Surgery — Patients will undergo metabolic surgery
  Arms: Metabolic Surgery

SUMMARY:
It is a prospective randomized trial on 218 subjects, 109 for each arms. The purpose of this trial is to compare very low calorie diet and metabolic surgery induced weight loss and its maintenance.

DETAILED DESCRIPTION:
Obesity is a leading public health issued associated with poor quality of life, morbidity and an increased mortality rate. Although metabolic surgery results in a greater weight loss when compared to non-surgical approaches, a low calorie diet associated with intensive maintenance session may be a valid alternative for weight loss. Since lifestyle interventions are safer and potentially more cost effective than metabolic surgery, this trial will test whether an intensive lifestyle intervention is as effective as metabolic surgery to induce weight loss and its maintenance.

A total of 218 participants will be randomly assigned to metabolic surgery (109) or intensive lifestyle intervention (109).

Clinical outcomes will be assessed at 25% reduction in Body Mass Index (BMI), at 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 69 years
* Body Mass Index ≥35 kg/m2 and at least one or more obesity-related co-morbidities such as type II diabetes (T2DM), hypertension, sleep apnea and other respiratory disorders, non-alcoholic fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease
* Body Mass Index ≥40 kg/m2

Exclusion Criteria:

* Pregnancy
* Active cancer
* End stage renal failure
* End stage liver failure
* Being unable to understand and sign informed consent

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to achieve a 25% reduction in Body Mass Index | 1-12 months

SECONDARY OUTCOMES:
Percentage of participants who achieve 25% reduction in Body Mass Index | 1-12 months
Time to achieve 25% reduction in Body Mass Index | 1-24months
Change in body composition (lean mass-all tissues in the body except bone and fat-fat mass, bone density and visceral fat) using dual energy X-ray absorptiometry (DXA), from baseline, at 25% weight loss, at 12 months follow up and at 24 months follow up | 1-24months
Change in glycated hemoglobin (HbA1c), from baseline, at 12 and 24 months follow up (patients with diabetes) | 1-24months
Change in fasting glucose and fasting insulin, from baseline, at 12 and 24 months follow up | 1-24months
Change in insulin resistance (assessed by HOMA-IR), from baseline, at 12 and 24 months follow up | 1-24months
Change in blood pressure, from baseline, at 12 and 24 months follow up | 1-24months
Change in total, HDL, LDL and total cholesterol from baseline, at 12 and 24 months follow up | 1-24months
Change in triglycerides from baseline, at 12 and 24 months follow up | 1-24months
Percentage of participants who maintain weight loss at 24 months follow up | 1-24months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University School of Medicine, Rome, Italy